CLINICAL TRIAL: NCT05988398
Title: Rigorous Evaluation of the READY to Stand Curriculum as a Tool to Prevent the Commercial Sexual Exploitation of Children Among Racially and Ethnically Diverse Urban Youth (PHASE II: OPEN PILOT TRIAL)
Brief Title: Preventing Commercial Sexual Exploitation of Children
Acronym: Project LIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska Lincoln (Other)
Collaborators: The Set Me Free Project (Unknown); Des Moines Public Schools (Unknown); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 22811; 1U01CE003405 (NIH)
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Results first posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Sex Trafficking; Sex Crimes; Commercial Sex; Sexual Violence; Child Abuse, Sexual; Sex Offense
Keywords: Human Trafficking; Sex Trafficking; Sex Crimes; Commercial Sex; Commercial Sexual Exploitation of Children; Prevention
MeSH Terms: conditions — Sex Work; Coitus

STUDY DESIGN:
Intervention Model Description: Two Schools will receive the intervention in addition to pre- and post- surveys. There is no control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RTS Intervention (Experimental): RTS intervention will include a total of one 120-minute session of programming delivered to school personnel, and six, 45-minute sessions (total = 4.5 hours) for students. There are five components in this intervention that both students and school personnels will receive: 1) Psychoeducation on CSEC, 2) Healthy relationship skills training, 3) Programming components to enhance valuing of self and others, 4) Bystander intervention skills, and 5) Social norms for both students and school personnel. Students will additionally receive programming on Identification of safe people and resources, while school personnel will receive programming on Responding to Student Disclosures, and Cultural Humility.
  Interventions: Behavioral: READY To Stand Curriculum

INTERVENTIONS:
Behavioral: READY To Stand Curriculum — Students will receive the RTS programming over six consecutive school days, spread over two weeks. The program is delivered in mixed-gender groups of 20 to 40 students and includes videos, small and large group discussions, activities, worksheets, and ample opportunities for skill-building. This curriculum is intended to be one piece of comprehensive prevention strategies that has the potential to make immediate and sustained impacts on reducing rates of CSEC perpetration in the lives of youth, including those most vulnerable to this pernicious crime.
  Other Names: RTS

SUMMARY:
The overall goal of the 5-year project is to conduct both a process and rigorous outcome evaluation of The Set Me Free Projects (SMFP) READY to Stand (RTS) curriculum with an eye toward widespread dissemination to other U.S. communities, if deemed effective.

DETAILED DESCRIPTION:
Detailed Description: The commercial sexual exploitation of children (CSEC) is a public health crisis in the U.S.1-4 Research has documented risk and protective factors across the social ecology for CSEC,2,5-8 that many perpetrators (traffickers, clients, recruiters) of CSEC are peers (e.g., romantic partners) 9-11 and adolescents report opportunities to intervene in situations of peer victimization (although not necessarily specific to CSEC).12-14 Prevention efforts with adolescents that seek to (1) reduce risk for CSEC perpetration; (2) reduce risk for CSEC victimization; and (3) increase positive bystander intervention in situations of CSEC is urgently needed. Thus, the goal of this multi-stakeholder collaboration-that includes researchers, educators, practitioners, and youth-is to conduct both a process and rigorous outcome evaluation of The Set Me Free Project's© (SMFP) READY to Stand (RTS)© curriculum-with an eye toward widespread dissemination to other U.S. communities, if deemed effective. This project is responsive to Research Priority Area 4 (preventing CSEC as a form of CSA) of RFA-CE-22-003. The implementation site includes eight high schools in Des Moines Public Schools (DMPS); students (naïve to the RTS curriculum) are largely racial/ethnic minority (65%) and low-income (76%). DMPS leadership have expressed a growing concern about the CSEC in their district and are eager to partner with researchers to rigorously evaluate the RTS curriculum. The RTS curriculum includes four, 45-minute modules implemented to high school students in mixed gender groups of ~25 students and provides students with psychoeducation on CSEC, healthy relationship skills training, identification of safe people/resources, and programming components to enhance valuing of self and others. As part of the proposed project, the RTS curriculum will be enhanced with two additional 45-minute modules on bystander intervention training in situations of CSEC and shifting school norms to be intolerant of all forms of violence, including CSEC. Additionally, school personnel participate in an enhanced (from 90 minutes to 120 minutes) training to equip them with skills to effectively respond to students' disclosures of CSEC and to reinforce programming messages. The RTS curriculum may also reduce other forms of violence such as teen dating violence (TDV) given it addresses risk and protective factors for multiple forms of violence. Despite its potential for reducing CSEC, the RTS curriculum has never been evaluated. Specific Aims are as follows: Refinement and Planning Phase (Component A): Convene a Research Advisory Board (RAB) that includes researchers, practitioners, educators, caregivers, and youth who will provide input on all research components of the project (Aim 1a). Conduct focus groups with students (n=80) and school personnel (n=60) to inform the refinement of the RTS curriculum and research procedures for Component B (Aim 1b). Enhance the existing RTS program manual and create a training manual to ensure consistent implementation, produce training manuals for use in subsequent clinical trials and dissemination, and develop fidelity measures (Aim 1c). Develop via cognitive interviews (n=20 youth, n=10 school personnel) and surveys (n=878) with students valid, reliable, and developmentally appropriate measures of CSEC perpetration, CSEC victimization, and CSEC bystander opportunity/action to be used in subsequent research, including Component B (Aim 1d). Conduct an open pilot trial of the RTS curriculum in one of the five traditional high schools and one of the three alternative schools in DMPS with students (n=878) and school personnel (n=78) to gain experience with the recruitment and assessment procedures and administration of the intervention; assess acceptability and safety of the research protocols; document initial trends, effect sizes, and CSEC incidence rates; and refine the intervention and research procedures in preparation for Component B (Aim 1e). Apply for additional funding under Component B and disseminate findings to diverse audiences in collaboration with the RAB (Aim 1f). All procedures for Component B will be ready for implementation by the end of Component A funding. Rigorous Evaluation Phase (Component B): Conduct a quasi-experimental study in which four traditional high schools in DMPS and two alternative high schools (not including the two high schools that participated in Component A) are demographically matched and randomly assigned to treatment or wait-list control conditions. Students (n=7,241) will complete baseline and 6-, 12-, and 18-month follow-up surveys to test the hypothesis that participation in the RTS program will lead to reductions in CSEC perpetration (primary outcome), as well as reductions in CSEC victimization and TDV and sexual violence victimization and perpetration and increases in bystander intervention in CSEC situations compared to participants in the waitlist control condition (secondary outcomes) (Aim 2a). We will assess mediators and demographic moderators of program impact (Aim 2b). Document via program observations of student and school personnel programming (Aim 2c), post-session surveys (n=7,241 students; n=396 school personnel) (Aim 2d), and post-program implementation key informant and stakeholder interviews (n=40: program facilitators [n=10], students [n=20], school personnel [n=10]) (Aim 2e) variations in implementation, unanticipated challenges, lessons learned, and perceptions of program impact. Determine costs associated with the program implementation (both student and school personnel programming) to inform future economic evaluation of the RTS curriculum (Aim 2f). Refine and assess validity and reliability of school personnel's' CSEC prevention related knowledge, attitudes, and skills (Aim 1g). Examine the preliminary impact of the RTS school personnel training curriculum on CSEC prevention related knowledge, attitudes, and skills as well as acceptability and perceptions of impact (Aim 1h).

ELIGIBILITY:
Inclusion Criteria:

* For school personnel, participants must be 18 years of age or older and currently employed at Hoover or All Points for the OPT and one of the eight high schools in DMPS for the survey development portion of the study (Aim 1g). We will include anyone working in administration (e.g., principal), teaching (e.g., academic subject matter instructor) or support service (e.g., counselor) capacity within any of the eight high schools encompassed within Des Moines Public School (DMPS) system.
* For students, participants must be in Grades 9 through 12 at one of the eight participating high schools in DMPS and be able to understand spoken English. For the OPT (Aims 1e, 1h) this includes Hoover and All Points.

Exclusion Criteria:

* For school personnel, not being 18 or older or currently employed at Hoover or All Points for the OPT and one of the eight high schools in DMPS.
* For students, being in Grades younger than 9 or older than 12 and not being enrolled in participating high school in DMPS.

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 356 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-05-29 (Actual); Study Completion 2024-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katie M Edwards, PhD, Principal Investigator — University of Nebraska Lincoln; Rochelle Dalla, PhD, Study Director — University of Nebraska Lincoln; Lorey Wheeler, PhD, Study Director — University of Nebraska Lincoln
Locations (1):
- [a school district in the Midwest], Des Moines, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
The level of public access will be restricted such that the data set will be available under certain use restrictions. More specifically, the PI intends to share the aggregated, de-identified quantitative survey data if users commit to the following: (a) using the data only for research purposes and not to identify any individual participant; (b) securing the data using appropriate computer technology; and (c) destroying or returning the data after analyses are completed. If the researcher agrees, in writing, to these stipulations, the PI will send the approved researcher the dataset prepared using SPSS 27.0 (or the latest version available). The prepared data set will not include identifying information about participants, schools, or DMPS. Research participants will be identified by number. Schools will be coded as a number so as not to identify the participating schools/district.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be made available likely around summer 2025. It will be made available indefinitely.
Access Criteria: See above in Plan Description

REFERENCES:
- [Background] Prevention CfDCa. Rigorously Evaluating Programs and Policies to Prevent Child Sexual Abuse (CSA) RFA-CE-22-003. 2021
- [Background] Anderson PM, Coyle KK, Johnson A, Denner J. An exploratory study of adolescent pimping relationships. J Prim Prev. 2014 Apr;35(2):113-7. doi: 10.1007/s10935-014-0338-3. PMID 24445410
- [Background] American Association of University Women Educational Foundation. Hostile hallways: Bullying, teasing, and sexual harassment in school. ERIC; 2001.
- [Background] Bal M. A Review of Human Dignity. Dignity in the Workplace. 2017:41-66.
- [Background] Bowers EP, Li Y, Kiely MK, Brittian A, Lerner JV, Lerner RM. The Five Cs model of positive youth development: a longitudinal analysis of confirmatory factor structure and measurement invariance. J Youth Adolesc. 2010 Jul;39(7):720-35. doi: 10.1007/s10964-010-9530-9. Epub 2010 Apr 16. PMID 20397040
- [Background] Centers for Disease Control and Prevention. 2019 Youth Risk Behavior Surveillance System results. U.S. Department of Health & Human Services. https://www.cdc.gov/healthyyouth/data/yrbs/index.htm
- [Background] Cook-Craig PG, Coker AL, Clear ER, Garcia LS, Bush HM, Brancato CJ, Williams CM, Fisher BS. Challenge and opportunity in evaluating a diffusion-based active bystanding prevention program: Green Dot in high schools. Violence Against Women. 2014 Oct;20(10):1179-202. doi: 10.1177/1077801214551288. Epub 2014 Sep 24. PMID 25255794
- [Background] Edwards KM, Banyard VL, Kirkner A. Parents Matter: A Descriptive Study of Parental Discussions With Teens About Violence Prevention and Related Topics. J Interpers Violence. 2022 Apr;37(7-8):NP3856-NP3874. doi: 10.1177/0886260520949153. Epub 2020 Aug 26. PMID 32842824
- [Background] Edwards KM, Banyard VL, Waterman EA, Mitchell KJ, Jones LM, Kollar LMM, Hopfauf S, Simon B. Evaluating the Impact of a Youth-Led Sexual Violence Prevention Program: Youth Leadership Retreat Outcomes. Prev Sci. 2022 Nov;23(8):1379-1393. doi: 10.1007/s11121-022-01343-x. Epub 2022 Mar 18. PMID 35303249
- [Background] Edwards KM, Littleton H. Development and pilot evaluation of an online intervention to prevent dating violence and problem drinking in sexual minority youth. University of Nebraska Lincoln, Lincoln, NE: National Institute of Health; 2021-2023.
- [Background] Edwards KM, Sessarego SN, Stanley LR, Mitchell KJ, Eckstein RP, Rodenhizer KAE, Leyva PC, Banyard VL. Development and Psychometrics of Instruments to Assess School Personnel's Bystander Action in Situations of Teen Relationship Abuse and Sexual Assault. J Interpers Violence. 2021 Feb;36(3-4):NP1586-1606NP. doi: 10.1177/0886260517746946. Epub 2017 Dec 20. PMID 29295034
- [Background] Franchino-Olsen H, Martin SL, Halpern CT, Preisser JS, Zimmer C, Shanahan M. Adolescent Experiences of Violence Victimizations Among Minors Who Exchange Sex/Experience Minor Sex Trafficking. J Interpers Violence. 2022 Sep;37(17-18):NP16277-NP16301. doi: 10.1177/08862605211021967. Epub 2021 Jun 30. PMID 34192962
- [Background] Hulsey L, Zief, S., & Murphy, L. PREP Entry and Exit Survey Measures Guide. 2022. https://www.prepeval.com/DataCollection/50273%20Data%20Dictionary%202022.pdf
- [Background] Jenkins N, Saiz C. The communication skills test. Unpublished manuscript, University of Denver, Denver, CO. 1995
- [Background] Johnson JG, Harris ES, Spitzer RL, Williams JB. The patient health questionnaire for adolescents: validation of an instrument for the assessment of mental disorders among adolescent primary care patients. J Adolesc Health. 2002 Mar;30(3):196-204. doi: 10.1016/s1054-139x(01)00333-0. PMID 11869927
- [Background] Lebech M. What is human dignity? Maynooth philosophical papers. 2004;2:59-69.
- [Background] Lerner, R. M., Almerigi, J. B., Theokas, C., & Lerner, J. V. (2005). Positive youth development a view of the issues. The journal of early adolescence, 25(1), 10-16.
- [Background] Monitoring the future national survey results on drug use, 1975-2020: Overview, key findings on adolescent drug use. https://eric.ed.gov/?id=ED611736.
- [Background] Park N. Character strengths and positive youth development. Annals of the American Academy of Political and Social Science. 2004;591(1):40-54. doi:10.1177/0002716203260079
- [Background] Proctor E, Silmere H, Raghavan R, Hovmand P, Aarons G, Bunger A, Griffey R, Hensley M. Outcomes for implementation research: conceptual distinctions, measurement challenges, and research agenda. Adm Policy Ment Health. 2011 Mar;38(2):65-76. doi: 10.1007/s10488-010-0319-7. PMID 20957426
- [Background] Project P. COMPREHENSIVE HUMAN TRAFFICKING ASSESSMENT. 2011
- [Background] Project SMF. READY to Stand Curriculum. 2021
- [Background] Quinn-Nilas C, Milhausen RR, Breuer R, Bailey J, Pavlou M, DiClemente RJ, Wingood GM. Validation of the Sexual Communication Self-Efficacy Scale. Health Educ Behav. 2016 Apr;43(2):165-71. doi: 10.1177/1090198115598986. Epub 2015 Aug 17. PMID 26286296
- [Background] Quirk, K., Newcomb, M. E., & Mustanski, B. (2018). LGBQ identity integration and the association with justification of violence. Psychology of Violence, 8(2), 184.
- [Background] Rothman EF, Paruk J, Cuevas CA, Temple JR, Gonzales K. The Development of the Measure of Adolescent Relationship Harassment and Abuse (MARSHA): Input From Black and Multiracial, Latinx, Native American, and LGBTQ+ Youth. J Interpers Violence. 2022 Mar;37(5-6):2126-2149. doi: 10.1177/0886260520936367. Epub 2020 Jul 5. PMID 32627640
- [Background] Waterman EA, Banyard VL, Edwards KM, Mauer VA. Youth perceptions of prevention norms and peer violence perpetration and victimization: A prospective analysis. Aggress Behav. 2022 Jul;48(4):402-417. doi: 10.1002/ab.22024. Epub 2022 Feb 16. PMID 35174509
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Ziebertz H-G, Döhnert S, Unser A. Predictors of attitudes towards human dignity: An empirical analysis among youth in Germany. Religion and civil human rights in empirical perspective. Springer; 2018:17-60.

RESULTS

PARTICIPANT FLOW:
Groups:
- RTS Intervention-School Personnel: RTS intervention will include a total of one 120-minute session of programming delivered to school personnel. There are five components in this intervention that school personnel will receive: 1) Psychoeducation on CSEC, 2) Healthy relationship skills training, 3) Programming components to enhance valuing of self and others, 4) Bystander intervention skills, and 5) Social norms for both students and school personnel. Students will additionally receive programming on Identification of safe people and resources, while school personnel will receive programming on Responding to Student Disclosures, and Cultural Humility.
- RTS Intervention-Students: RTS intervention will include six, 45-minute sessions (total = 4.5 hours) for students. There are five components in this intervention that students will receive: 1) Psychoeducation on CSEC, 2) Healthy relationship skills training, 3) Programming components to enhance valuing of self and others, 4) Bystander intervention skills, and 5) Social norms for both students and school personnel. Students will additionally receive programming on Identification of safe people and resources, while school personnel will receive programming on Responding to Student Disclosures, and Cultural Humility.
  READY To Stand Curriculum: Students will receive the RTS programming over six consecutive school days, spread over two weeks. The program is delivered in mixed-gender groups of 20 to 40 students and includes videos, small and large group discussions, activities, worksheets, and ample opportunities for skill-building. This curriculum is intended to be one piece of comprehensive prevention strategies that has the potential to make immediate and sustained impacts on reducing rates of CSEC perpetration in the lives of youth, including those most vulnerable to this pernicious crime.
Period: Overall Study
Arm/Group | RTS Intervention-School Personnel | RTS Intervention-Students
Started | 68 | 212
Completed | 47 | 107
Not Completed | 21 | 105
Not completed — Lack of time | 21 | 0
Not completed — Absent from school | 0 | 38
Not completed — Chose not to participate | 0 | 42
Not completed — Other commitments (e.g., sports) | 0 | 25

BASELINE CHARACTERISTICS:
Population: School personnel from all high schools within the district were invited to complete the survey. Total of 68 school personnel attended the workshop and completed the feedback form. From two public Midwestern high schools (one traditional and one alternative), a total of 229 students consented to participate, with a final sample of 177 students who completed the survey.
Groups:
- Total: Total of all reporting groups
Arm/Group | RTS Intervention-School Personnel | RTS Intervention-Students | Total
Number analyzed (Participants) | 68 | 177 | 245
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5714 (11.28582) | 15.93 (1.62) | 28.03 (15.70)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Row population differs from overall due to missing values. RTS Intervention - Student group didn't have the option for "Other" as a gender
  Participants
    Man | 5 | 74 | 79
    Woman | 20 | 79 | 99
    Other | 0 | 19 | 19
    Declined to answer or Unknown | 43 | 5 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 35 | 39
  Not Hispanic or Latino | 22 | 126 | 148
  Unknown or Not Reported | 42 | 16 | 58
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 23 | 23
  Native Hawaiian or Other Pacific Islander | 0 | 3 | 3
  Black or African American | 1 | 64 | 65
  White | 22 | 51 | 73
  More than one race | 0 | 19 | 19
  Unknown or Not Reported | 45 | 16 | 61

OUTCOME MEASURES:

1. Primary Outcome: Commercial Sexual Exploitation Children (CSEC) Perpetration (STUDENT Reported)
Description: For the initial pool of items, we identified existing CSEC perpetration items from The National Study on Adolescent to Adult Health (ADD Health; Franchino-Olsen et al., 2021) and The My Life My Choices evaluation study (Rothman et al., 2021). The scale consists of 21 statements and response options included yes, no, or I do not want to answer this question. A total score is calculated from the sum of the items, with higher scores reflective of a higher sex trafficking perpetration experiences in the past month.
Time Frame: 1-month post RTS delivery
Population: Students from two public Midwestern high schools (one traditional and one alternative)
Measure: Count of Participants; unit: Participants
Arm/Group | RTS Intervention-Students
Number analyzed (Participants) | 107
Participants
  No | 79
  Yes | 11
  Declined to answer or Unknown | 17

2. Secondary Outcome: Commercial Sexual Exploitation of Children (CSEC) Victimization (STUDENT Reported)
Description: For the initial pool of items, we identified existing CSEC victimization items from The National Study on Adolescent to Adult Health (ADD Health; Franchino-Olsen et al., 2021) and The My Life My Choices evaluation study (Rothman et al., 2021). The scale consists of 21 statements and response options included yes, no, or I do not want to answer this question. A total score is calculated from the sum of the items, with higher scores reflective of a higher sex trafficking victimization experiences in the past month.
Time Frame: One-month post RTS delivery
Population: Students from two public Midwestern high schools (one traditional and one alternative)
Measure: Count of Participants; unit: Participants
Arm/Group | RTS Intervention-Students
Number analyzed (Participants) | 107
Participants
  No | 12
  Yes | 6
  Declined to answer or Unknown | 89

3. Secondary Outcome: Bystander Readiness to Help (STUDENT Reported)
Description: The bystander readiness to help scale was based on the denial subscale of the readiness to help scale (D-RHS; Banyard et al., 2014) to assess students's awareness of and willingness to engage in prevention efforts regarding CSE among high school students in their school district. These items have similarly been adapted for measuring opinions regarding relationship abuse and/or sexual assault among high school students (Edwards et al., 2018). The scale consists of four statements using a 4-point Likert scale (1 = strongly agree to 4 = strongly disagree). A total score is calculated from the average of the items, with higher scores reflective of a greater sense of need and the willingness to engage.
Time Frame: One-month post RTS delivery
Population: Students from two public Midwestern high schools (one traditional and one alternative)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RTS Intervention-Students
Number analyzed (Participants) | 107
score on a scale | 2.7857 (0.54988)

4. Secondary Outcome: Sexual Assault Victimization (STUDENT Reported)
Description: Behaviorally worded items to assess students' self-reports of experiencing past month sexual assault victimization, with items adapted from Cook-Craig et al. (2014). The scale consists of 4 items with response options (1=Yes, 0=No, and -999=I don't want to answer). The original scale has response options ranging from 0-4 (0=0 times, 4=10+ times). A total score is calculated from taking a count of items with a response of "yes", with scores ranging from 0-4. Higher scores indicate more instances of sexual assault victimization having occurred.
Time Frame: 1-month post RTS delivery
Population: Students from two public Midwestern high schools (one traditional and one alternative)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RTS Intervention-Students
Number analyzed (Participants) | 107
score on a scale | 0.0833 (0.3814)

5. Secondary Outcome: Sexual Assault Perpetration (STUDENT Reported)
Description: Behaviorally worded items to assess students' self-reports of experiencing past month sexual assault perpetration, with items adapted from Cook-Craig et al. (2014). The scale consists of 4 items with response options (1=Yes, 0=No, and -999=I don't want to answer). The original scale has response options ranging from 0-4 (0=0 times, 4=10+ times). A total score is calculated from taking a count of items with a response of "yes", with scores ranging from 0-4. Higher scores indicate more instances of sexual assault perpetration having occurred.
Time Frame: One-month post RTS delivery
Population: Students from two public Midwestern high schools (one traditional and one alternative)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RTS Intervention-Students
Number analyzed (Participants) | 107
score on a scale | 0.0333 (0.1810)

6. Secondary Outcome: Sexual Harassment Victimization (STUDENT Reported)
Description: Behaviorally worded items to assess past month students' self-reports of experiencing sexual harassment victimization. Items adapted from American Association of University Women Educational Foundation (2001, p.21). The scale consists of 2 items with response options (1=Yes, 0=No, and -999=I don't want to answer). A total score is calculated from taking a count of items with a response of "yes", with scores ranging from 0-2. Higher scores indicate more instances of sexual harrassment victimization having occurred.
Time Frame: 1-month post RTS delivery
Population: Students from two public Midwestern high schools (one traditional and one alternative)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RTS Intervention-Students
Number analyzed (Participants) | 107
score on a scale | 0.4677 (0.6457)

7. Secondary Outcome: Sexual Harassment Perpetration (STUDENT Reported)
Description: Behaviorally worded items to assess past month students' self-reports of experiencing sexual harassment perpetration. Items adapted from American Association of University Women Educational Foundation (2001, p.21). The scale consists of 2 items with response options (1=Yes, 0=No, and -999=I don't want to answer). A total score is calculated from taking a count of items with a response of "yes", with scores ranging from 0-2. Higher scores indicate more instances of sexual harrassment perpetration having occurred.
Time Frame: 1-month post RTS delivery
Population: Students from two public Midwestern high schools (one traditional and one alternative)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RTS Intervention-Students
Number analyzed (Participants) | 107
score on a scale | 0.1774 (0.4625)

8. Secondary Outcome: Stalking Victimization (STUDENT Reported)
Description: Behaviorally worded items to assess students' past month self-reports of experiencing stalking victimization, with items adapted from(Cook-Craig et al. 2014). The scale consists of 3 items with response options (1=Yes, 0=No, and -999=I don't want to answer). The original scale has response options ranging from 0-4 (0=0 times, 4=10+ times). A total score is calculated from taking a count of items with a response of "yes", with scores ranging from 0-3. Higher scores indicate more instances of stalking victimization having occurred.
Time Frame: 1-month post RTS delivery
Population: Students from two public Midwestern high schools (one traditional and one alternative)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RTS Intervention-Students
Number analyzed (Participants) | 107
score on a scale | 0.3115 (0.6962)

9. Secondary Outcome: Stalking Perpetration (STUDENT Reported)
Description: Behaviorally worded items to assess students' past month self-reports of experiencing stalking perpetration, with items adapted from(Cook-Craig et al. 2014). The scale consists of 3 items with response options (1=Yes, 0=No, and -999=I don't want to answer). The original scale has response options ranging from 0-4 (0=0 times, 4=10+ times). A total score is calculated from taking a count of items with a response of "yes", with scores ranging from 0-3. Higher scores indicate more instances of stalking perpetration having occurred.
Time Frame: 1-month post RTS delivery
Population: Students from two public Midwestern high schools (one traditional and one alternative)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RTS Intervention-Students
Number analyzed (Participants) | 107
score on a scale | 0.1833 (0.53652)

10. Secondary Outcome: Dating Violence Victimization (STUDENT Reported)
Description: The Measure of Adolescent Relationship Harassment and Abuse (MARSHA; Rothman et al. 2020) was used to assess past month dating violence victimization. The scale consists of two subscales, Physical abuse (7 items) and Isolation (3 items), with response options of 1=Yes, 0=No, and -999=I don't want to answer. A total score is calculated from the counting the nunber of items answers as "yes". Higher scores indicate more instances of dating violence victimization having occurred.
Time Frame: 1-month post RTS delivery
Population: Students from two public Midwestern high schools (one traditional and one alternative)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RTS Intervention-Students
Number analyzed (Participants) | 107
score on a scale | 0.4286 (1.27904)

11. Secondary Outcome: Dating Violence Perpetration (STUDENT Reported)
Description: The Measure of Adolescent Relationship Harassment and Abuse (MARSHA; Rothman et al. 2020) was used to assess past month dating violence perpetration. The scale consists of two subscales, Physical abuse (7 items) and Isolation (3 items), with response options of 1=Yes, 0=No, and -999=I don't want to answer. A total score is calculated from the counting the nunber of items answers as "yes". Higher scores indicate more instances of dating violence perpetration having occurred.
Time Frame: 1-month post RTS delivery
Population: Students from two public Midwestern high schools (one traditional and one alternative)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RTS Intervention-Students
Number analyzed (Participants) | 107
score on a scale | 0.1429 (0.35274)

12. Secondary Outcome: Youth Violence (STUDENT Reported)
Description: The Youth Risk Behavior Surveillance System (YRBS; Centers for Disease Control and Prevention, 2019) was used to measure past month physical fights, fear of going to school, and weapon carrying. The scale consisted of 4 items with response options of 1=Yes, 0=No, and -999=I don't want to answer. A total score is calculated from the counting the nunber of items answers as "yes". Higher scores indicate more instances of youth violence having occurred.
Time Frame: 1-month post RTS delivery
Population: Students from two public Midwestern high schools (one traditional and one alternative)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RTS Intervention-Students
Number analyzed (Participants) | 107
score on a scale | 0.1833 (0.50394)

13. Secondary Outcome: Depression (STUDENT Reported)
Description: The Patient Health Questionnaire (PHQ-9) modified (Johnson et al. 2002) was used to measure past two week depression. The scale consisted of 8 items with response options from Not at all (0) to Nearly every day (3) and I don't want to answer (-999). The toal score is calculated from the average of the items, with higher scores representing higher depression symptoms.
Time Frame: 1-month post RTS delivery
Population: Students from two public Midwestern high schools (one traditional and one alternative)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RTS Intervention-Students
Number analyzed (Participants) | 107
score on a scale | 1.0342 (0.84775)

14. Secondary Outcome: Academic & Career Commitment (STUDENT Reported)
Description: Items from Hulsey et al. (2022) were used to measures students intentions on graduating high school/getting a GED as well as having a job/career. The scale consisted of 5 items with response scales from Not at all true of me (1) to Extremely true of me (4) and I don't want to answer this question (-999). The total scores were calculated from the average of the items, with higher scores representing higher academic and career commitment.
Time Frame: 1-month post RTS delivery
Population: Students from two public Midwestern high schools (one traditional and one alternative)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RTS Intervention-Students
Number analyzed (Participants) | 107
score on a scale | 2.8762 (0.6024)

15. Other Pre Specified Outcome: CSEC Knowledge (STUDENT Reported)
Description: Consistent with other measures of sexual violence/teen dating violence knowledge for youth (Edwards et al., 2019), questions (e.g., "most victims are trafficked by strangers") are True/False. We provide youth a definition of CSE, specifically, sex trafficking. We created six items to measure adolescents' knowledge of CSE. The respondents are asked if they believe the statements to be true or false. Items are scored based upon whether they were answered correctly (1) or incorrectly (0). The scores were then averaged to create a cumulative score that reflects the proportion of statements answered correctly (Min=0, Max=6).
Time Frame: 1-month post RTS delivery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RTS Intervention-Students
Number analyzed (Participants) | 107
score on a scale | 0.8711 (0.2001)

16. Other Pre Specified Outcome: Efficacy (STUDENT Reported)
Description: Author created items to assess confidence in resistance to being a victim of CSEC. Two statements asked how confident the participant is in recognizing sex trafficking (i.e., "If someone tried to force you into sex trafficking, how confident are you that you would recognize it?"), and keeping it from happening (i.e., "If someone tried to force you into sex trafficking, how confident are you that you would be able to keep it from happening?"). Participants rated the statements using the four options: Not at all confident (1), Somewhat confident (2), Very confident (3) , and I don't want to answer this question (-999). Total score was calculated into a mean with higher scores indicating higher efficacy.
Time Frame: 1-month post RTS delivery
Population: Students from two public Midwestern high schools (one traditional and one alternative)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RTS Intervention-Students
Number analyzed (Participants) | 107
score on a scale
  Recognizing Sex Trafficking | 2.47 (0.66)
  Keeping it from Happening | 2.37 (0.72)

17. Other Pre Specified Outcome: Valuing Self (STUDENT Reported)
Description: The Valuing of Self (e.g., "I have value") scales was adapted from measures and conceptualizations of positive youth development (PYD; Bowers et al., 2010; Lerner et al., 2005; Park, 2010) and dignity scales (Bal, 2017; Lebech, 2004; Ziebertz et al., 2018). Prior to the questions, a definition of value was provided. The scale included eight statements. Participants rated statements from strongly disagree (1) to strongly agree (4). Scores were calculated by taking the average of the items with higher scores indicating higher sense of valuing of self.
Time Frame: 1-month post RTS delivery
Population: Students from two public Midwestern high schools (one traditional and one alternative)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RTS Intervention-Students
Number analyzed (Participants) | 107
score on a scale | 3.2432 (0.57972)

18. Other Pre Specified Outcome: Valuing Other(STUDENT Reported)
Description: The Valuing of Others (e.g., "All people have value") scale was adapted from measures and conceptualizations of positive youth development (PYD; Bowers et al., 2010; Lerner et al., 2005; Park, 2010) and dignity scales (Bal, 2017; Lebech, 2004; Ziebertz et al., 2018). Prior to the questions, a definition of value was provided. The scale included eight statements. Participants rated statements from strongly disagree (1) to strongly agree (4). Scores were calculated by taking the average of the items with higher scores indicating higher sense of valuing of other.
Time Frame: 1-month post RTS delivery
Population: Students from two public Midwestern high schools (one traditional and one alternative)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RTS Intervention-Students
Number analyzed (Participants) | 107
score on a scale | 3.1601 (0.60016)

19. Other Pre Specified Outcome: Perceptions of Social Norms of Prevention of CSEC (STUDENT Reported)
Description: The Social Norms scale (Waterman et al., 2022) (adapted from prior work; Waterman et al., 2022) is composed of four subscales that gauges personal beliefs, perceptions of friends, perceptions of other high school students in this district, and perceptions of school personnel in the district regarding their beliefs on sex trafficking. Participants rated all statements on a scale from strongly disagree (1) to strongly agree (4). An option of I don't want to answer was also provided. Subscale scores were calculated from the average of the items, with higher scores representing social norms less supporting of sex trafficking, including personal beliefs, perceptions of friends, other high school students, and school personnel.
Time Frame: 1-month post RTS delivery
Population: Students from two public Midwestern high schools (one traditional and one alternative)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RTS Intervention-Students
Number analyzed (Participants) | 107
score on a scale
  Personal Beliefs | 3.4063 (0.5248)
  Perceptions of Friends | 3.1908 (0.59479)
  Percceptions of HS Students in their district | 3.0784 (0.66649)
  Perceptions of School Personnel in their district | 3.4286 (0.65544)

20. Other Pre Specified Outcome: Prevention-related Communication With School Personnel (STUDENT Reported)
Description: We adapted items created by Edwards et al. (2021, 2022). The eight statements focused on things school personnel had discussed with students, including general items such as how to have healthy relationships and their futures, as well as CSE items, including sex trafficking, sexual assault, and dating and/or domestic violence, and to what extent they agreed with each statement (1 = strongly disagree to 4 = strongly agree). The final score was the average of the scale items, with higher values indicating more engagement between students and school personnel.
Time Frame: 1-month post RTS delivery
Population: Students from two public Midwestern high schools (one traditional and one alternative)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RTS Intervention-Students
Number analyzed (Participants) | 107
score on a scale | 2.8483 (0.55481)

21. Other Pre Specified Outcome: CSEC Knowledge (SCHOOL PERSONNEL Reported)
Description: Consistent with other measures of sexual violence/teen dating violence knowledge for youth (Edwards et al., 2019), questions (e.g., "most victims are trafficked by strangers") are True/False. We provide youth a definition of CSE, specifically, sex trafficking. We created nine items to assess school personnel's general knowledge about CSE and the roles school personnel can play in its prevention. The respondents are asked if they believe the statements to be true or false. Items are scored based upon whether they were answered correctly (1) or incorrectly (0). The scores were then averaged to create a cumulative score that reflects the proportion of statements answered correctly
Time Frame: 1-month post RTS delivery
Population: School Personnel from all high schools within the district
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RTS Intervention-School Personnel
Number analyzed (Participants) | 47
score on a scale | 0.947 (0.067)

22. Other Pre Specified Outcome: Bystander Readiness to Help (SCHOOL PERSONNEL Reported)
Description: The bystander readiness to help scale was based on the denial subscale of the readiness to help scale (D-RHS; Banyard et al., 2014b) to assess school personnel's awareness of and willingness to engage in prevention efforts regarding CSE among high school students in their school district. These items have similarly been adapted for measuring opinions regarding relationship abuse and/or sexual assault among high school students (Edwards et al., 2018). The scale consists of four statements using a 4-point Likert scale (1 = strongly agree to 4 = strongly disagree). A total score is calculated from the average of the items, with higher scores reflective of a greater sense of need and the willingness to engage.
Time Frame: 1-month post RTS delivery
Population: School Personnel from all high schools within the district
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RTS Intervention-School Personnel
Number analyzed (Participants) | 47
score on a scale | 3.379 (0.412)

23. Other Pre Specified Outcome: Perceptions of Social Norms of Prevention of CSEC (SCHOOL PERSONNEL Reported)
Description: The Social Norms scale (Waterman et al., 2022) (adapted from prior work; Waterman et al., 2022) is composed of four subscales that gauges personal beliefs, perceptions of friends, perceptions of other high school students in this district, and perceptions of school personnel in the district regarding their beliefs on sex trafficking. For school personnels, three out of the four subscales were included (i.e., personal belief, perceptions of high school students in this district, and perceptions of school personnel in the district). Participants rated all statements on a scale from strongly disagree (1) to strongly agree (4). An option of I don't want to answer was also provided. Subscale scores were calculated from the average of the items, with higher scores representing social norms less supporting of sex trafficking, including personal beliefs, other high school students, and school personnel.
Time Frame: 1-month post RTS delivery
Population: School Personnel from all high schools within the district
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RTS Intervention-School Personnel
Number analyzed (Participants) | 47
score on a scale
  Personal Beliefs | 3.74375 (0.520378)
  Perceptions of Students | 2.923611 (0.492150)
  Perceptions of School Personnel | 3.618421 (0.502483)

24. Other Pre Specified Outcome: Prevention-related Communication With School Personnel (SCHOOL PERSONNEL Reported)
Description: as for outcome 20
Time Frame: 1-month post RTS delivery
Population: School Personnel from all high schools within the district
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RTS Intervention-School Personnel
Number analyzed (Participants) | 47
score on a scale | 3.28 (0.501)

25. Other Pre Specified Outcome: Cultural Humility (SCHOOL PERSONNEL Reported)
Description: The Cultural Humility scale was based on The Multicultural Teaching Competency Scales (Spanierman et al., 2011). The scale consists of 16 statements using a 5-point Likert scale (1 = strongly disagree to 5 =strongly agree). The total score is calculated from the average of the items, with higher scores reflective of a higher sense of cultural humility.
Time Frame: 1-month post RTS delivery
Population: School Personnel from all high schools within the district
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RTS Intervention-School Personnel
Number analyzed (Participants) | 47
score on a scale | 4.0444 (0.5901)

ADVERSE EVENTS:
Time Frame: Data on adverse events were collected throughout the study from baseline survey (1 week before programming), during intervention (6 days of programming), post-program survey (1-month follow-up from program end).
Description: All-Cause Mortality is not a possible outcome of this trial.
Arm/Group | RTS Intervention-School Personnel | RTS Intervention-Students
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/212
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/212
Other Adverse Events (participants affected / at risk) | 0/68 | 212/212
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RTS Intervention-School Personnel (N=68) | RTS Intervention-Students (N=212)
Content Delivery (Social circumstances) | 0 (0) | 212 (212) — School educators who were also project partners were selected to deliver the youth curriculum, but due to an oversight had not yet received approval from the IRB before delivering the curriculum in school.
Recruitment (Social circumstances) | 0 (0) | 0 (0) — Staff members were recruiting participants and conducting outreach visits in the community going door-to-door using a door knocking protocol that had not yet been approved in this study but had been previously used in other studies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-11-09): https://cdn.clinicaltrials.gov/large-docs/98/NCT05988398/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-20): https://cdn.clinicaltrials.gov/large-docs/98/NCT05988398/SAP_003.pdf
  • Informed Consent Form (2024-04-02): https://cdn.clinicaltrials.gov/large-docs/98/NCT05988398/ICF_002.pdf